CLINICAL TRIAL: NCT01685164
Title: The Effect of Uterine Size and Posture on Intrauterine Contraception in Nulliparous Women
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Satu P. Suhonen, MD, PhD, Physician in chief, Centralized Family Planning, City of Helsinki Health Centre, Helsinki University Central Hospital
Other Study IDs: 1491/13/03/03/2010
Record Dates: First submitted 2012-08-30; First posted 2012-09-14 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Intrauterine Contraception
Keywords: nulliparous; IUD; IUS; insertion; expulsion
MeSH Terms: interventions — Posture; High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- LNG-IUS: Nulliparous women
  Interventions: Other: Evaluation of uterine size and posture with ultrasound, IUD insertion, one year follow-up.
- Cu-IUD: Nulliparous women
  Interventions: Other: Evaluation of uterine size and posture with ultrasound, IUD insertion, one year follow-up.

INTERVENTIONS:
Other: Evaluation of uterine size and posture with ultrasound, IUD insertion, one year follow-up. — Evaluation of uterine size and posture with ultrasound, IUD insertion, one year follow-up.

SUMMARY:
As intrauterine contraception is an increasingly popular form of contraception the objective of our study is to examine if uterine size or posture affects the insertion or use of intrauterine devices. Nulliparous women requesting either the levonorgestrel-releasing device (LNG-IUS) or a copper-IUD (NovaT) are recruited and followed for one year.

DETAILED DESCRIPTION:
Prospective observational study among nulliparous women requesting intrauterine contraception.

ELIGIBILITY:
Inclusion Criteria:

- nulliparous women with no previous history of IUD use

Exclusion Criteria:

* malformation of uterus
* myomas
* acute gynecological infection
* malignant uterine or cervical tumor

In addition if requesting a Cu-IUD

* heavy menstruations
* iron deficiency
* bleeding disorder
* copper allergy or Wilson's disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of nulliparous women attending the centralized Family planning center of the City of Helsinki requesting intrauterine contraception, either the LNG-IUS or a Cu-IUD.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The effect of uterine size or posture on IUD insertion. | Day 1
  The size of the uterine cavity (cm) and the flexion angle of the uterus are determined at insertion using ultrasonography. This is compared with assessment of perception of insertion pain both by the patient and the inserting doctor is evaluated as well as the easiness if insertion (by the doctor).

SECONDARY OUTCOMES:
Satisfaction and continuation rate with intrauterine contraception. | 3 months
  Clinical evaluation including gynecological examination is at 3 months after insertion. Patterns of bleeding and severeness of pain are followed daily for the 90 first days after insertion.
Satisfaction and continuation rate with intrauterine contraception. | 12 months
  A second clinical evaluation including gynecological examination is at 12 months after insertion. Patterns of bleeding and severeness of pain are followed daily for the last 90 days of the first year of use of intrauterine contraception.

CONTACTS AND LOCATIONS:
Locations (1):
- Contraceptive unit of city of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Kaislasuo J, Heikinheimo O, Lahteenmaki P, Suhonen S. Menstrual characteristics and ultrasonographic uterine cavity measurements predict bleeding and pain in nulligravid women using intrauterine contraception. Hum Reprod. 2015 Jul;30(7):1580-8. doi: 10.1093/humrep/dev102. Epub 2015 May 19. PMID 25990577
- [Derived] Kaislasuo J, Heikinheimo O, Lahteenmaki P, Suhonen S. Predicting painful or difficult intrauterine device insertion in nulligravid women. Obstet Gynecol. 2014 Aug;124(2 Pt 1):345-353. doi: 10.1097/AOG.0000000000000362. PMID 25004340